CLINICAL TRIAL: NCT06635603
Title: HYPERTENSIVE CRISIS AND ATMOSPHERIC PRESSURE RELATIONSHIP: A PROSPECTIVE STUDY
Brief Title: HYPERTENSIVE CRISIS AND ATMOSPHERIC PRESSURE RELATIONSHIP
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Etimesgut Military Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Hypertension, ATM pressure
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Hypertensive Urgency; Weather
Keywords: atmospheric pressure; hypertension; hypertensive urgency
MeSH Terms: conditions — Hypertensive Crisis; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hypertension: patients admitted to emergency department with grade 3 (systolic ≥180 and/or diastolic ≥110 mmHg) blood pressure

SUMMARY:
relationship between the onset times of symptoms and the regions of patients presenting to the emergency department with hypertensive crisis (systolic ≥180 and/or diastolic ≥110 mmHg) and the fluctuations in atmospheric pressure

DETAILED DESCRIPTION:
Hypertensive emergency is defined as grade 3 hypertension (systolic ≥180 and/or diastolic ≥110 mmHg) that causes end-organ damage, requiring urgent intervention and intensive care admission . Hypertensive crisis is described as severe hypertension not associated with end-organ damage. Some sources define hypertensive crisis as hypertension of grade 3 or higher, while others refer to it as severe hypertension without specifying a threshold .

Literature reviews, published guidelines, and studies indicate that the definitions and treatment approaches for hypertensive crisis differ between Europe and America, with variations in management from one physician to another . Seasonal blood pressure fluctuations are influenced by external temperature, indoor temperature, humidity, atmospheric pressure, and wind . Notably, during periods of low atmospheric pressure, blood pressure measurements show statistically significant increases compared to other days . Consequently, the frequency of life-threatening conditions associated with hypertension, such as intracranial hemorrhage and abdominal aortic aneurysm rupture, has been observed to increase on days when atmospheric pressure changes .

In our study, we aim to investigate the relationship between the onset times of symptoms and the regions of patients presenting to the emergency department with hypertensive crisis (systolic ≥180 and/or diastolic ≥110 mmHg) and the fluctuations in atmospheric pressure

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above
2. Hypertensive crisis (systolic ≥180 and/or diastolic ≥110 mmHg)

Exclusion Criteria:

1. Patients presenting with hypertensive emergency (those with end-organ damage)
2. Patients who have traveled to another city or district within the last 4 days
3. Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to emergency department with hypertensive urgency ( systolic ≥180 and/or diastolic ≥110 mmHg )
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Hypertensive Crisis | from enrollment to the end of follow up duration of 7 days
  Patients' blood pressure values evaluation in terms of atmospheric pressure and weather conditions

CONTACTS AND LOCATIONS:
Overall Officials: Gulsen AKCAY, ass. prof., Study Director — Ankara Etlik City Hospital
Locations (1):
- Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salvetti M, Paini A, Colonetti E, Tarozzi L, Bertacchini F, Aggiusti C, Stassaldi D, Rosei CA, Rosei EA, Muiesan ML. Hypertensive emergencies and urgencies: a single-centre experience in Northern Italy 2008-2015. J Hypertens. 2020 Jan;38(1):52-58. doi: 10.1097/HJH.0000000000002213. PMID 31415308
- [Result] Jehn M, Appel LJ, Sacks FM, Miller ER 3rd; DASH Collaborative Research Group. The effect of ambient temperature and barometric pressure on ambulatory blood pressure variability. Am J Hypertens. 2002 Nov;15(11):941-5. doi: 10.1016/s0895-7061(02)02999-0. PMID 12441212
- [Result] Modesti PA, Morabito M, Massetti L, Rapi S, Orlandini S, Mancia G, Gensini GF, Parati G. Seasonal blood pressure changes: an independent relationship with temperature and daylight hours. Hypertension. 2013 Apr;61(4):908-14. doi: 10.1161/HYPERTENSIONAHA.111.00315. Epub 2013 Feb 4. PMID 23381792